CLINICAL TRIAL: NCT05934643
Title: An Observational Cohort Study to Assess the Postoperative Physical Activity of Patients Undergoing Elective Colorectal Resection.
Brief Title: An Observational Cohort Study to Assess the Postop Activity of Colorectal Patients Undergoing Elective Surgery (PHYSPAL)
Acronym: PHYSPAL
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 23025
Record Dates: First submitted 2023-06-09; First posted 2023-07-07 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-04

CONDITIONS: Colorectal (Colon or Rectal) Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — 4-amino-4'-hydroxylaminodiphenylsulfone; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ActivPAL accelerometer — All patient will have an accelerometer (activPAL) applied to characterise the type and quantity of movement during the inpatient postoperative period after undergoing major surgery for colorectal cancer surgery.
Other: Hospital Anxiety and Depression Scale (HADS) Questionnaire — The use of the HADS questionnaire to ascertain if any correlation between level of activity and and inpatient mood.

SUMMARY:
All participants will have a physical activity monitor placed onto the right thigh in the midline which will start collecting data at midnight on the first postoperative day. This will continue until discharge or day 7, whichever is earlier. This is a non-invasive measure of activity and can discriminate between whether a patient is lying, sitting, standing or walking. There is no control group.

DETAILED DESCRIPTION:
Recruited patients from the colorectal clinic at the Royal Derby Hospital will be invited to be included in the study, and can either attend the University of Nottingham, Centre Of Metabolism, Ageing & Physiology (COMAP) research group unit at the Royal Derby Hospital Centre or discuss the trial in detail over the phone after which a consent form will be sent to them (either by post or email). If they agree to inclusion in the study the consent form will be brought with them to be completed on the day of surgery. On the morning of surgery they will have their consent recorded and the activPAL™ accelerometer applied to the anterior thigh.

The activPAL™ is a non-invasive physical monitor that records periods spent, lying, walking and engaging in more strenuous activity. This will remain in situ for 7 days, or until discharge, whichever comes first. The investigators will ask participants to complete a short diary to note down any times the monitor is removed and the time of sleep and waking. After removal - the data is uploaded (it does not include any person-identifiable data) for analysis using software on a local computer in the COMAP unit. After discharge, they will have 2 x telephone calls and/or emails at day 10 and at day 28 to follow up from the research team to monitor progress for the next 30 days. If they develop any complications including readmission data within that time period, this will be collected from the participants' notes along with demographic data and postoperative pathology and recorded. Complications will be graded as per the Clavien-Dindo Classification system.

On postoperative day 3, day 5 and day 7 (if still an inpatient) they will also be asked to complete the Hospital Anxiety and Depression Scale (HADS) paper questionnaire. Just prior to discharge, they will complete the discharge questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and over
* Clinical diagnosis of colorectal cancer due to undergo surgical resection with curative intent
* Must be able to give informed consent

Exclusion Criteria:

* Lacking capacity to consent
* Undergoing emergency surgery
* Undergoing defunctioning surgery prior to neoadjuvant treatment
* Undergoing surgery with palliative intent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting to Royal Derby Hospital who have gone through colorectal multidisciplinary team (MDT) meeting with a plan for surgical resection of colorectal cancer with curative intent.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Average daily energy expenditure in MET.h | 30 days from operation date
  Using the ActivPAL accelerometers, to assess the MET.h per each postoperative day

SECONDARY OUTCOMES:
Step count | From the first postoperative day until discharge or day 7, whichever is sooner.
  Using the ActivPAL accelerometers, record average daily step count
Sit to stands | From the first postoperative day until discharge or day 7, whichever is sooner.
  Using the ActivPAL accelerometers, record average daily sit-to-stand count
Time spent in bed | From the first postoperative day until discharge or day 7, whichever is sooner.
  Using the ActivPAL accelerometers, record average time spent in bed in hours.
30-day complication rate | 30 days from operation date.
  All postoperative complications will be recorded and classified as per the Clavien-Dindo classification.

CONTACTS AND LOCATIONS:
Overall Officials: Jon Lund, DM, FRCS, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Royal Derby Hospital, Derby, United Kingdom

IPD SHARING:
Plan to Share IPD: No